CLINICAL TRIAL: NCT04310384
Title: A Randomized Cross-Over Trial to Determine Whether the 'ShuttleScope® Laryngoscope is Inferior, Equal or Superior Compaired to Macintosh Laryngoscope to Perform Successful Endotracheal Intubation in a Manikin Model.
Brief Title: 'Single Hand Used inTubaTing Laryngoscope Evaluation' Study
Acronym: SHUTTLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Jose Medrano Laporte, MD PhD, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2019/259
Record Dates: First submitted 2020-03-05; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Respiratory Failure; Cardiac Arrest; Difficult Intubation; Anesthesia Intubation Complication
Keywords: Airway management; Videolaryngoscope; Mannequin; Endotracheal Intubation
MeSH Terms: conditions — Respiratory Insufficiency; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endotracheal Intubation, gold standart (Active Comparator): Standart of Care with Macintosh laryngoscope
  Interventions: Device: MacIntosh Laryngoscope
- Alternative (Active Comparator): Endotracheal Intubation with novel device
  Interventions: Device: ShuttleScope

INTERVENTIONS:
Device: ShuttleScope — Alternative intervention
  Arms: Alternative
Device: MacIntosh Laryngoscope — Gold Standart
  Arms: Endotracheal Intubation, gold standart

SUMMARY:
This is a study to compare the new ShuttleScope with the standard Macintosh Laryngoscope

DETAILED DESCRIPTION:
Following a 5 minutes workshop with an instructor structured demonstration and practice with both devices, the participants attempt intubation in a normal airway scenario with the Macintosh Laryngoscope and the novel ShuttleScope®, in a manikin model.

ELIGIBILITY:
Inclusion Criteria:

* Medecine students from the Basque Country University (UPV/EHU)

Exclusion Criteria:

* Other operators different from the ones described above
* Previous experience with ShuttleScope videolaryngoscope
* informed consent non available

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Success Rate | During intubation time, intubation attempts allows maximum 3 times, within 90 sec in each time
  Number of succesfull intubations after three attempts
Time to Endotracheal Intubation | During intubation time, intubation attempts allows maximum 3 times, within 90 sec in each time
  The duration of intubation is defined as the time from inserting videolaryngoscope, intubating a tube, to withdrawing videolaryngoscope using a stopwatch.

SECONDARY OUTCOMES:
Incidence of' oesophageal intubation | During intubation time, intubation attempts allows maximum 3 times, within 90 sec in each time
  Number of oesophageal Intubations after three attempts
Ease of insertion | During intubation time, intubation attempts allows maximum 3 times, within 90 sec in each time ]
  Described by the operator and defined in a subjective visual analogue scale (VAS) from 0 to 10 for each of the devices (0 extremely difficult to 10 extremely easy)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Miguel Alonso Babarro, Principal Investigator — Airwaymedicalinnovations
Locations (1):
- Hospital Virtual, Unidad Docente de Medicina, Facultad de Medicina y Enfermeria de la Universidad del País Vasco (UPV/EHU), Vitoria-Gasteiz, Alava, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Airwaymedicalinnovations — https://airwaymedicalinnovations.com/